CLINICAL TRIAL: NCT01936844
Title: Interleukin-1 Blockade in Acute Decompensated Heart Failure
Brief Title: Interleukin (IL)-1 Blockade in Acute Heart Failure (Anakinra ADHF)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCU HM15347
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anakinra (short) (Experimental): Anakinra 100 mg twice daily for the first 3 days followed by 100 mg daily for days 4-14
  Interventions: Drug: Anakinra (high dose); Drug: Anakinra (standard dose)
- Placebo (Placebo Comparator): Placebo injections twice daily for the first 3 days then once daily for days 4-14.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra (high dose) — Anakinra 100 mg daily twice daily for days 1, 2, and 3
  Arms: Anakinra (short)
Drug: Anakinra (standard dose) — Anakinra 100 mg daily for days 4-14
  Arms: Anakinra (short)
Drug: Placebo — Placebo twice daily for days 1, 2, and 3
  Arms: Placebo
Drug: Placebo — Placebo daily for days 4-14
  Arms: Placebo

SUMMARY:
Anakinra ADHF is a double-blind randomized clinical trial of anakinra, recombinant human interleukin-1 receptor blocker, or placebo in patients with acute decompensated heart failure with the aim to quench the acute inflammatory response, as measured by the area-under-the-curve for C reactive protein over 14 days.

ELIGIBILITY:
Inclusion Criteria:

All 5 criteria need to be met for enrollment of the patient in the study

1. Primary diagnosis of acute decompensated heart failure within the last 24 hours as evidenced by both of the following:

   1. dyspnea or respiratory distress or tachypnea at rest or with minimal exertion
   2. evidence of elevated cardiac filling pressure or pulmonary congestion (at least one of the conditions must be met);

   i. pulmonary congestion/edema at physical exam OR chest x-ray; ii. plasma Brain Natriuretic Peptide (BNP) levels ≥200 pg/mL; iii.invasive measurement of left ventricular end-diastolic pressure >18 mmHg or of pulmonary artery occluding pressure (wedge) >16 mmHg.
2. Left ventricular systolic dysfunction (LVEF<40%) during index hospitalization or prior 12 months.
3. Age ≥18 years old
4. Willing and able to provide written informed consent.
5. Screening plasma C-reactive protein levels >5 mg/L.

Exclusion Criteria Subjects will not be eligible if they meet any of the following 15 exclusion criteria.

1. The primary diagnosis for admission is NOT decompensated heart failure, including diagnosis of acute coronary syndromes, hypertensive urgency/emergency, tachy- or brady-arrhythmias.
2. Concomitant clinically significant comorbidities that would interfere with the execution or interpretation of the study including but not limited to acute coronary syndromes, uncontrolled hypertension or orthostatic hypotension, tachy- or brady-arrhythmias, acute or chronic pulmonary disease or neuromuscular disorders affecting respiration.
3. Recent (previous 3 months) or planned cardiac resynchronization therapy (CRT), coronary artery revascularization procedures, or heart valve surgeries.
4. Previous or planned implantation of left ventricular assist devices or heart-transplant.
5. Chronic use of intravenous inotropes.
6. Recent (<14 days) use of immunosuppressive or anti-inflammatory drugs (not including Non-Steroidal Anti-Inflammatory Drugs [NSAIDs]).
7. Chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus).
8. Active infection (of any type);
9. Chronic/recurrent infectious disease (including Hepatitis B virus [HBV], Hepatitis C virus [HCV], and HIV/AIDS).
10. Prior (within the past 10 years) or current malignancy.
11. Any comorbidity limiting survival or ability to complete the study.
12. End stage kidney disease requiring renal replacement therapy.
13. Neutropenia (<2,000/mm3) or Thrombocytopenia (<50,000/mm3).
14. Pregnancy.
15. Angina, arrhythmias, or electrocardiograph (ECG) changes that limit maximum exertion during cardiopulmonary exercise testing obtained during the baseline testing.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Data may be available upon request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra (Short) | Placebo
Started | 15 | 15
Completed | 9 | 8
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra (Short) | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [49 to 64] | 54 [49 to 66] | 58 [49 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
C-reactive protein [Median (Inter-Quartile Range); unit: mg/L] | 22.3 [10.8 to 95.9] | 27.4 [12.0 to 47.2] | 23.8 [10.9 to 46.9]

OUTCOME MEASURES:

1. Primary Outcome: C Reactive Protein
Description: The proportional area-under-the-curve for plasma C reactive protein (CRP) levels measured during the first 3 days of admission. The proportion (y-axis) is calculated at each time-point with respect to the baseline CRP. The resultant y-axis is a unitless proportion. The x-axis is listed as "days"
Time Frame: 3 days
Population: 1 patient in each group withdrew from the study prior to collection of data for the primary endpoint.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Anakinra (Short) | Placebo
Number analyzed (Participants) | 14 | 14
days | 2.09 [1.73 to 2.61] | 2.93 [2.36 to 3.79]

2. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Change in left ventricular ejection fraction (LVEF) between admission and 14 day follow up. This value is expressed as absolute change in measured LVEF. For example, if baseline LVEF = 20% and 14 day LVEF = 25%, this would be reported as an absolute change of 5%.
Time Frame: 14 days
Population: Some patients did not undergo LVEF assessment at 14 days because they did not show up to their scheduled appointment.
Measure: Median (Inter-Quartile Range); unit: percent LVEF
Arm/Group | Anakinra (Short) | Placebo
Number analyzed (Participants) | 7 | 7
percent LVEF | 10 [3 to 14] | 0 [-16 to 5]

3. Secondary Outcome: Brachial Artery Vasoreactivity
Description: Change in flow mediated vasodilatation (FMD) of the brachial artery. Brachial artery FMD is calculated as the percentage increase in brachial artery diameter with hyperemia (an increase in the quantity of blood flow to a body part) induced relative to the resting brachial artery diameter. Percentage of brachial artery diameter is measured as FMD diameter/basal diameter. The change is FMD is reported as the % change in FMD from baseline to 14 days.
Time Frame: 14 days
Population: Some patients did not undergo assessment at 14 days because they did not show up to their scheduled appointment.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Anakinra (Short) | Placebo
Number analyzed (Participants) | 8 | 7
percentage change | 41.7 [-44.5 to 98.2] | -45.2 [-101.0 to 45.8]

ADVERSE EVENTS:
Arm/Group | Anakinra (Short) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/15 | 4/15
Other Adverse Events (participants affected / at risk) | 4/15 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (Short) (N=15) | Placebo (N=15)
Worsening heart failure or Readmission for heart failure (Cardiac disorders) | 2 (2) | 3 (3)
Serious infection/sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (Short) (N=15) | Placebo (N=15)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No